CLINICAL TRIAL: NCT06433323
Title: Evaluation of Biological Anti-aging Efficacy of the Cosmetic Night Cream RV4983A- LA3365 in Women After 2 Months of Daily Use
Brief Title: Biological Anti-aging Efficacy of a Cosmetic Night Cream
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Collaborators: SpinControl (Unknown)
Responsible Party: Sponsor
Other Study IDs: RV4983A20240122
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treated group : Healthy female adults
  Interventions: Other: Anti-aging cosmetic care product

INTERVENTIONS:
Other: Anti-aging cosmetic care product — This is an intra-individual comparison study.
  * frequency of application: Once a day (in the evening)
  * modalities of application: Apply the cream on the tested area determined by the randomization
  * duration of investigational product application: 56 days (a window of + 72 hours is allowed)

SUMMARY:
In a previous study, the cosmetic night cream RV4983A- LA3365 has proven a great efficacy in reducing the clinical signs of skin aging, as well as a great tolerance. The skin structure and composition greatly evolve over the time, and deciphering the biological mechanisms by which the cosmetic night cream RV4983A- LA3365 reduces the signs of skin aging is therefore of great interest to deepen our efficacy evaluation and knowledge on skin aging biology.

DETAILED DESCRIPTION:
An intra-individual, comparative study randomized will be conducted as monocentric trial in female adult

46 subjects are included

4 visits are planned:

* Visit 1 (D1): Inclusion and 1st product application
* Visit 2 (D28): Phone call follow-up
* Visit 3 (D57): End of application and biopsies
* Visit 4 (7 days after V3): Biopsies control and end-of-study

For a subject completing the study, the theoretical investigational product application will be 56 consecutive days up to 59 days maximum.

The maximal duration of participation for a subject is 68 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject with phototype I, II or III according to the Fitzpatrick scale

Non-inclusion Criteria:

* Criteria related to the subject's health / skin :

  * Subject having any dermatologic condition or characteristics (like tattoo) on any of the target areas liable to interfere with the study assessments
  * Subject having a dermatological condition, an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the Investigator hazardous for the subject or incompatible with the study requirements
  * Subject having received on any of target areas artificial UV exposure, excessive or prolonged exposure to natural sunlight within 2 weeks before the inclusion visit or planning to be exposed to artificial UV, excessive or prolonged natural sunlight during the study and up to 3 months after completion of study participation
  * Subject hirsute on the target areas
  * Subject having contraindication to the local anaesthetic used for biopsies
  * Subject with known immune deficiency
  * Subject with a recognised addiction to alcohol or drug
  * Subject with a scar pathology or pathology with consequences for healing such as diabetes
  * Subject with known history of hepatitis B or C or known HIV positive status
  * Subject with hereditary or acquired haemostasis disorder
  * Smoker > 10 cigarettes/day with nicotine (or equivalent in electronic cigarettes)
* Criteria related to treatments and/or products:

  * Surgical, chemical or significant invasive treatment on any of the target areas within 6 months before the inclusion or planned during the study
  * Techniques with aesthetic aim on any of the target areas (laser, pulsed flash lamp etc.) or injections of reshaping products (collagen, hyaluronic acid, botulinic toxin etc.) within 6 months before the inclusion or planned during the study
  * Oral isotretinoin taken within 6 months before the inclusion or planned during the study
  * Phototherapy treatment on any of the target areas within 2 months before the inclusion or planned during the study
  * Systemic treatment likely to affect haemostasis (anticoagulants, platelet antiaggregants, etc.) taken within the weeks before the inclusion or planned during the study
  * Systemic treatment may interfere with the healing process (non-steroidal anti-inflammatory drugs, corticosteroids, immunosuppressants) taken within the weeks before the inclusion or planned during the study
  * Systemic treatment or topical treatment applied on any target areas likely to interfere with the local anesthetic (anti-arhythmic, beta blockers etc.) within the weeks before the inclusion or planned during the study
  * Topical non-steroidal anti-inflammatory, dermocorticoids, immunomodulators applied on any of the target areas within the 2 weeks before the inclusion or planned during the study
  * Topical skincare product (e.g. exfoliation, scrub, body mask) applied on any of the target areas within 7 days before the inclusion or planned during the study

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy female volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Biological efficacy assessed by the analysis of proteins expression related to aging. | Day 57
  Will be determined from skin biopsies.
General safety assessed by the occurence of Adverse Events. | Day 1 to Day 68
  The occurrence of Adverse Events will be determined by the subject's spontaneous reporting, the investigator's non-leading questioning and his/her clinical evaluation.
Compliance calculated from data reported by the subject in her diary. | Day 1 to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth GUITTON-OUDET, Dr, Principal Investigator — SpinControl
Locations (1):
- SpinControl, Tours, Indre et Loire, France

IPD SHARING:
Plan to Share IPD: No